CLINICAL TRIAL: NCT00997594
Title: Changes in Adrenal Hormones During Adrenal Radiofrequency Ablation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mie University (Other)
Responsible Party: Principal Investigator, Koichiro Yamakado, Clinical Professor, Mie University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 274; No secondary IDs
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Results first posted 2011-02-23 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Adrenal Tumors
Keywords: adrenal gland
MeSH Terms: conditions — Adrenal Gland Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adrenal radiofrquency (RF) ablation (Active Comparator): Patients who wll receive adrenal RF ablation.
  Interventions: Procedure: Radiofrequency ablation
- Abdominal RF ablation other than adrenal gland (Active Comparator): Patients who will receive abdominal radiofrequency ablation other than adrenal gland.
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — Radiofrequency (RF) ablation was done after RF electrodes were placed in the adrenal tumor in the adrenal RF ablation group. RF ablation was done after RF electrodes were placed in the targeted abdominal tumors other than adrenal gland in the abdominal RF ablation other than adrenal gland group.

SUMMARY:
The purpose of this study is to evaluate changes in adrenal hormones during adrenal radiofrequency (RF) ablation.

DETAILED DESCRIPTION:
Adrenal radiofrequency (RF) ablation has been increasingly used for the treatment of unresectable adrenal tumors. But one of the major complication is a increase in blood pressure. Hormonal release during RF ablation is considered the cause of hypertension. But there has been no evidence that adrenal hormones affects changes in blood pressure. In this prospective study, we evaluate the changes in adrenal hormones during RF ablation and clarify the cause of hypertensive crisis.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable adrenal tumor which will be treated by radiofrequency (RF)ablation
* Blood pressure is 140mmHg or less before RF ablation
* Age of 20-years or more
* Performance status of 0 or 1
* Agreement from the patient

Exclusion Criteria:

* Platelet count of 50,000/mm^3 or International normalized ratio (INR)>1.5

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koichiro Yamakado, MD, Study Chair — Mie University School of Medicine
Locations (2):
- Japan (2):
  - Mie University Hospital, Tsu, Mie-ken
  - Mie University, Tsu, Mie-ken

RESULTS

PARTICIPANT FLOW:
Groups:
- Adrenal Radiofrequency Ablation: Patients who received adrenal radiofrequency (RF) ablation.
- Abdominal Radiofrequency Ablation Other Than Adrenal Gland: Patients who received radiofrequency (RF) ablation other than adrenal gland such as liver and kidney.
Period: Overall Study
Arm/Group | Adrenal Radiofrequency Ablation | Abdominal Radiofrequency Ablation Other Than Adrenal Gland
Started | 9 | 9
Completion of Ablation Procedure | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adrenal Radiofrequency Ablation | Abdominal Radiofrequency Ablation Other Than Adrenal Gland | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 3 | 11
  >=65 years | 1 | 6 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (13) | 71 (12) | 65 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  Japan | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Increase in Catecholamine
Time Frame: One day
Reporting Status: Not Posted

2. Secondary Outcome: Increase in Cortisol
Time Frame: 1 day
Reporting Status: Not Posted

3. Primary Outcome: Serum Cathecholamine Levels
Time Frame: around one year
Reporting Status: Not Posted, anticipated posting 2015-10
Measure: Mean

4. Primary Outcome: Number of Participants With Hypertension During Adrenal or Non-adrenal Radiofrequency Ablation
Description: Blood pressure was monitored during radiofrequency (RF) ablation. The frequency of hypertension (systolic blood pressure of more than 200 mmHg) was evaluated and compared between the adrenal and non-adrenal (RF ablation other than adrenal gland) RF ablation groups.
Time Frame: 1 week
Measure: Number; unit: participants
Arm/Group | Adrenal Radiofrequency Ablation | Abdominal Radiofrequency Ablation Other Than Adrenal Gland
Number analyzed (Participants) | 9 | 9
participants | 6 | 1
Statistical Analysis 1: Comparison: Adrenal Radiofrequency Ablation vs Abdominal Radiofrequency Ablation Other Than Adrenal Gland; Test type: Non-Inferiority or Equivalence — Just a comparison of the percentage of hypertension between the 2 patient groups; p < 0.05, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: 1 week to 1 year (mean, 215 days)
Arm/Group | Adrenal Radiofrequency Ablation | Abdominal Radiofrequency Ablation Other Than Adrenal Gland
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

LIMITATIONS AND CAVEATS:
Small patient series is one of limitations of this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes